CLINICAL TRIAL: NCT02766374
Title: Heart Rate Variability Biofeedback: It's Role in Asthma Therapeutics
Acronym: BioAce
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Wamboldt, MD (Other)
Collaborators: Rutgers University (Other); National Jewish Health (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Fred Wamboldt, MD, Executive Director Research Administration, National Jewish Health
Organization: National Jewish Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HL089495-01A2 (NIH); R01HL089495-01A2 (NIH)
Record Dates: First submitted 2014-02-14; First posted 2016-05-09 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Asthma; Biofeedback; Heart rate variability biofeedback; Inhaled corticosteroids
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart Rate Variability Biofeedback (Experimental): During the first training session, we will measure heart rate variability (HRV) amplitude while the patient breathes for two minutes at a frequency ranging between 4.5-6.5 breaths/min, providing a "pacing stimulus" for this purpose. In subsequent sessions, the individual will be given personal heart rate variability biofeedback (HRV-BF), and instructed to increase the amplitude of heart rate oscillations, using a cardiotachometer tracing and frequency peaks as biofeedback stimuli, while avoiding hyperventilation symptoms, by breathing more shallowly, although slowly, at whatever frequency produces maximum-amplitude HRV.
  Interventions: Behavioral: Heart rate variability biofeedback
- Placebo Biofeedback (Placebo Comparator): A credible Placebo Biofeedback (PBO-BF) consists of: 1) receiving EEG/music biofeedback (actually, a mildly relaxing intervention, using EEG biofeedback to alternately increase and decrease frontal/occipital EEG alpha rhythms while listening to relaxing music), and 2) listening to recorded sounds of nature along with relaxing music with instructions to maintain a condition of "relaxed alertness." For home training, subjects will be given "placebo" StressEraser programmed to give feedback to maintain their breathing at baseline rate.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback — Biofeedback teaches voluntary control of physiological functions by providing instantaneous feedback of variations in that bodily activity. Feedback usually is given in the form of visual and/or auditory signals derived from physiological recording devices. Among its salutary effects is a sense of medical self-efficacy, i.e., less dependency on medical professionals for maintaining personal health.
  The HRV-BF protocol we have developed and propose to examine herein works by a different pathway. It involves teaching the individual to increase the amplitude of heart rate accelerations during inhalation and de-celerations during exhalation, thus increasing the amplitude of respiratory sinus arrhythmia (RSA).
  Arms: Heart Rate Variability Biofeedback
Behavioral: Placebo — The method consists of: 1) receiving EEG/music biofeedback (actually, a mildly relaxing intervention, using EEG biofeedback to alternately increase and decrease frontal/occipital EEG alpha rhythms while listening to relaxing music), and 2) listening to recorded sounds of nature along with relaxing music with instructions to maintain a condition of "relaxed alertness." For home training, subjects will be given "placebo" StressEraser programmed to give feedback to maintain their breathing at baseline rate.
  Arms: Placebo Biofeedback

SUMMARY:
The goal of this research study to see whether biofeedback therapy helps treat asthma, and if so, how it works. Biofeedback is a treatment method that can teach how to bodily control. Biofeedback is widely used to help people relax. In this study however, the investigators want to learn if a specific type of biofeedback actually improves asthma in a way that might allow the reduction or elimination of other controller treatments like inhaled-corticosteroids.

DETAILED DESCRIPTION:
The purpose of this study is to determine the role of Heart rate variability biofeedback (HRV-BF) in asthma management as either a controller (alternative) or bronchodilator (complementary) treatment, with respect to the current treatment of choice, inhaled corticosteroid (ICS) therapy, using different methods from participants that demonstrated clinically significant improvement in asthma outcomes in the investigator's previous research (1), and adding a second site not involved in the investigator's previous work.

Inflammation of airways is viewed as the core pathophysiologic process in asthma. It is thought to render airways more reactive, and therefore, more susceptible to bronchoconstriction, leading to asthma exacerbations. Asthma is an episodic disease, where the goal of therapy is to reduce susceptibility to exacerbations, which may cause severe, even life-threatening illness. Anti-inflammatory medications reduce airways reactivity, while bronchodilator medications primarily relieve symptoms once an asthma exacerbation is in process, and may stop progressive constriction of airway smooth muscles (ASM). An anti-inflammatory effect of HRV-BF would have important implications for asthma management because adherence to ICS regimens is low due to a significant degree to feared side effects of prolonged steroid medication. Even if HRV-BF is found to only allow partial reduction in ICS requirements, this still would likely represent a major advance in asthma care.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate persistent asthma for at least the past one year
* Patients must not have taken oral or inhaled anti-inflammatory agents, including ICS and leukotriene inhibitors, for at least one month prior to study entry; and anti-IgE medications at least the past six months. Documented use of inhaled short-acting or long-acting β2-agonists during the month prior to study entry is, however, required. Xanthines, long-acting anticholinergics, and long-acting β2-agonists must be withdrawn within 72 hours upon entering the screening phase; short acting anticholinergics must be withdrawn within 48 hours before entering the screening phase. Patients will be required to abstain from these medications for the duration of study participation.
* FEV1 values must be ≥60% of predicted normal values following a 6 hour albuterol withhold, and reversibility of FEV1 of at least 12% (equal to or greater than 200 cc) following up to four puffs of albuterol must occur; or asthma physician at study site must state based on medical history, exam, and spirometry data that patient has presumptive mild-moderate persistent asthma.
* Lack of current asthma control as evidenced by ACT ≤ 19, or rescue use of B2-agonist ≥ 2/week within past 2 weeks, or waking due to asthma ≥ 1/week within past 2 weeks.
* Patients must be non-smokers for at least the past year and have less than a 15 pack-year smoking history. This will minimize the risk of co-occurring COPD
* Behavioral/linguistic competence: Ability to complete questionnaires and assessments in English
* Patients must give informed consent prior to any study procedures.

Exclusion Criteria:

* Diagnosis of severe persistent asthma
* 2 or more inpatient hospitalizations in the past year for asthma exacerbations;
* History of only seasonal asthma
* Patients with serious concomitant disease
* Patients who have had a respiratory tract infection within 4 weeks of screening
* Patients with a history of chronic bronchitis, COPD, or emphysema
* Patients with a history of alcohol or drug abuse, or emotional or cognitive problems requiring psychotropic medication or likely to interfere procedural and treatment adherence
* Any other clinically relevant deviation from normal in general medical history, physical examination, or laboratory parameters that would limit participation or interfere with study procedures and/or data collection;
* Presence of exclusive extra-thoracic airway dysfunction
* Women who are pregnant
* Presence of a heart rhythm or other abnormality of heart rhythm on screening EKG that could preclude ac-curate HRV assessment
* Chronically taking any medication likely to affect the autonomic or respiratory systems
* Asthma therapy and concomitant medication
* Previous participation in an investigational drug trial within 30 days prior to screening.
* Concurrent participation in any other clinical trial or observational study at any time in the study.
* Planning to move away from the area within the next 4 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-12; Primary Completion 2015-10 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick S Wamboldt, MD, Principal Investigator — National Jewish Health; Paul Lehrer, PhD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - Rutgers Robert Wood Johnson Medical School, Piscataway, New Jersey

REFERENCES:
- [Result] Lehrer PM, Irvin CG, Lu SE, Scardella A, Roehmheld-Hamm B, Aviles-Velez M, Graves J, Vaschillo EG, Vaschillo B, Hoyte F, Nelson H, Wamboldt FS. Heart Rate Variability Biofeedback Does Not Substitute for Asthma Steroid Controller Medication. Appl Psychophysiol Biofeedback. 2018 Mar;43(1):57-73. doi: 10.1007/s10484-017-9382-0. PMID 29124506

RESULTS

PARTICIPANT FLOW:
Groups:
- HRV Biofeedback: During the first training session, we will measure heart rate variability (HRV) amplitude while the patient breathes for two minutes at a frequency ranging between 4.5-6.5 breaths/min, providing a "pacing stimulus" for this purpose. In subsequent sessions, the individual will be given personal HRV biofeedback, and instructed to increase the amplitude of heart rate oscillations, using a cardiotachometer tracing and frequency peaks as biofeedback stimuli, while avoiding hyperventilation symptoms, by breathing more shallowly, although slowly, at whatever frequency produces maximum-amplitude HRV. This procedure detailed in Lehrer, P. M., Vaschillo, B., Zucker, T., Graves, J., Katsamanis, M.,Aviles, M., & Wamboldt, F. S. (2013). Protocol for heart rate variability biofeedback training. Biofeedback, 41(3), 98-109.
- EEG+ Biofeedback: Included instructions to increase and decrease EEG alpha from the right frontal to occipital areas (F4 to Oz), to listen regularly to relaxing music and to do paced breathing at the baseline rate of spontaneous breathing observed during a nondemanding task. Procedure detailed in Lehrer, P. M., Hochron, S. M., Mayne, T., Isenberg, S., Carlson, V., Lasoski, A. M., … Rausch, L. (1994). Relaxation and music therapies for asthma among patients prestabilized on asthma medication. Journal of Behavioral Medicine, 17(1), 1-24.
Period: Overall Study
Arm/Group | HRV Biofeedback | EEG+ Biofeedback
Started | 35 | 33
Completed | 25 | 30
Not Completed | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- HRV Biofeedback: Biofeedback to maximaize heart rate variability. Procedure detailed in Lehrer, P. M., Vaschillo, B., Zucker, T., Graves, J., Katsamanis, M.,Aviles, M., & Wamboldt, F. S. (2013). Protocol for heart rate variability biofeedback training. Biofeedback, 41(3), 98-109.
- Total: Total of all reporting groups
Arm/Group | HRV Biofeedback | EEG+ Biofeedback | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [26 to 45] | 31 [26 to 48] | 34 [26 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 31 | 25 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 17 | 21 | 38
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 4 | 0 | 4
Reported use of Short Acting Beta Adrenergic Medication (SABA) > 3/week [Count of Participants; unit: Participants] — SABA medication is used to treat asthma exacerbations, and using SABA > 3 times/week is taken as an indication of poorly controlled asthma.
  Participants | 3 | 7 | 10
Asthma Control Test (ACT) score total [Mean (Inter-Quartile Range); unit: units on a scale] — Range = 5-25 Scores > 19 indicate well-controlled asthma
  units on a scale | 20 [17.5 to 22.5] | 20 [16.6 to 23] | 20 [18 to 22]
Percent of Asthma Control Test (ACT) score ≤ 19 [Count of Participants; unit: Participants] — Range = 5-25 Scores > 19 indicate well-controlled asthma
  Participants | 18 | 20 | 38
Baseline provocative conc causing 20% fall in forced expiratory volume in 1 sec (PC20FEV1) (mg/ml) [Median (Inter-Quartile Range); unit: mg/ml] — Score represents the dose of methacholine that results in a 20% fall in Forced Expiratory Volume in 1 sec (FEV1). Doses start at 0.31 mg/ml and doubling doses of methacholine up to 25 mg/ml are given with test stopped once a ≥ 20% fall in FEV1 is achieved, with the result reported being the interpolated concentration of methacholine that produced a 20% drop. If a 20% was not achieved with the highest dose of methacholine (i.e., 25 mg/ml) a score of 25 is assigned.
  Range = 0.31-25 mg/ml
  mg/ml | 1.66 [1.10 to 5.0] | 1.40 [.51 to 3.35] | 1.46 [.79 to 5.0]
Forced Expiratory Volume in 1 sec (FEV1) (L) [Median (Inter-Quartile Range); unit: Liters (L)] — Quantity of air exhaled in the first second of a forced expiratory maneuver from maximum vital capacity measured using a spirometer.
  Liters (L) | 2.79 [2.20 to 3.19] | 3.01 [2.46 to 3.43] | 2.89 [2.24 to 3.36]
Precent predicted Forced Expiratory Volume in 1 sec (FEV1) [Median (Inter-Quartile Range); unit: Percent] — The percent predicted FEV1 is the FEV1 normalized as a percentage based on standards for an average healthy person of same age, race, height, and gender.
  Percent | 86.7 [68.7 to 97.9] | 84.1 [71.8 to 99.9] | 85.9 [71.0 to 98.0]
Forced Vital Capacity (FVC) (L) [Median (Inter-Quartile Range); unit: Liters (L)] — Total air exhaled in a forced expiratory maneuver from maximum vital capacity measured using a spirometer.
  Liters (L) | 3.78 [3.19 to 4.47] | 4.11 [3.42 to 4.98] | 4.04 [3.31 to 4.78]
Precent predicted Forced Vital Capacity (FVC) [Median (Inter-Quartile Range); unit: Percent] — The percent predicted FVC is the FVC normalized as a percentage based on standards for an average healthy person of same age, race, height, and gender.
  Percent | 102.2 [82.8 to 108.7] | 103.7 [90.0 to 109.8] | 103.0 [87.5 to 108.7]
Peak Expiratory Flow Rate (PEFR) (L/s) [Median (Inter-Quartile Range); unit: Liters/second (L/s)] — Peak expiratory flow rate during a forced airway maneuver from maximum vital capacity measured using a spirometer or a peak flow meter.
  Liters/second (L/s) | 6.90 [5.75 to 7.90] | 7.66 [6.26 to 9.14] | 7.27 [6.01 to 8.42]
Precent predicted Peak Expiratory Flow Rate (PEFR) [Median (Inter-Quartile Range); unit: Percent] — The percent predicted PEFR is the PEFR normalized as a percentage based on standards for an average healthy person of same age, race, height, and gender.
  Percent | 92.2 [80.7 to 99.9] | 92.6 [80.2 to 114.7] | 92.2 [80.7 to 107]
Exhaled Nitric Oxide cocentration (eNO) (ppb) [Median (Inter-Quartile Range); unit: parts per billion (p/b)] — Exhaled concentration of nitric oxide in parts per billion (eNO). eNO greater than 50 ppb indicates that eosinophilic inflammation of the airways is likely to be present and, in symptomatic patients, responsiveness to corticosteroid medications is likely.
  parts per billion (p/b) | 35.0 [20.0 to 61.0] | 43.0 [24.0 to 84.0] | 40.5 [21.0 to 71.0]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
  Scores = 25-29.9 indicate overweight status, Scores ≥ 30 indicate obese status
  kg/m^2 | 28.53 [24.78 to 31.65] | 27.41 [22.32 to 31.57] | 28.27 [22.93 to 31.57]

OUTCOME MEASURES:

1. Primary Outcome: Magnitude Change of Airway Reactivity Measured by Methacholine PC20FEV1
Description: Change in PEC20FEV1 measured after biofeedback from the PC20FEV1 measured at baseline
Time Frame: 4-weeks
Measure: Mean (95% Confidence Interval); unit: mg/ml
Groups:
- HRV-BF: During the first training session, we will measure heart rate variability biofeedback amplitude while the patient breathes for two minutes at a frequency ranging between 4.5-6.5 breaths/min, providing a "pacing stimulus" for this purpose. In subsequent sessions, the individual will be given personal HRV biofeedback, and instructed to increase the amplitude of heart rate oscillations, using a cardiotachometer tracing and frequency peaks as biofeedback stimuli, while avoiding hyperventilation symptoms, by breathing more shallowly, although slowly, at whatever frequency produces maximum-amplitude HRV.
- PBO-BF: The method consists of: 1) receiving EEG/music biofeedback (actually, a mildly relaxing intervention, using EEG biofeedback to alternately increase and decrease frontal/occipital EEG alpha rhythms while listening to relaxing music), and 2) listening to recorded sounds of nature along with relaxing music with instructions to maintain a condition of "relaxed alertness." For home training, subjects will be given "placebo" StressEraser programmed to give feedback to maintain their breathing at baseline rate.
Arm/Group | HRV-BF | PBO-BF
Number analyzed (Participants) | 35 | 33
mg/ml | 2.9782 [1.393 to 6.3675] | 2.1181 [1.2133 to 3.6977]
Statistical Analysis 1: Comparison: HRV-BF vs PBO-BF; Test type: Superiority; p > 0.1, GEE regression

ADVERSE EVENTS:
Time Frame: 4 week run-in, then 10 weeks of biofeedback.
Arm/Group | HRV Biofeedback | EEG+ Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes